CLINICAL TRIAL: NCT00953524
Title: Immunogenicity and Safety of Multiple Formulations of an A/H1N1 Pandemic Vaccine in Healthy Adult and Elderly Subjects
Brief Title: A Study of Different Formulations of an A/H1N1 Pandemic Vaccine in Healthy Adults and the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FUF14; UTN: U1111-1111-4798 (Other: WHO)
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza; Pandemic Flu; Swine-origin A/H1N1 Influenza; Adult
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A/H1N1 Vaccine Group 1 (Experimental): Participants will receive A/H1N1 vaccine formulation 1
  Interventions: Biological: Monovalent Subvirion A/H1N1 Influenza vaccine (7.5 µg of HA)
- A/H1N1 Vaccine Group 2 (Experimental): Participants will receive A/H1N1 vaccine formulation 2
  Interventions: Biological: Monovalent Subvirion A/H1N1 Influenza vaccine (15 µg of HA)
- A/H1N1 Vaccine Group 3 (Experimental): Participants will receive A/H1N1 Vaccine formulation 3
  Interventions: Biological: Monovalent Subvirion A/H1N1 Influenza vaccine (30 µg of HA)
- Placebo Group (Placebo Comparator): Participants will receive a placebo vaccine
  Interventions: Biological: Normal saline solution (placebo)

INTERVENTIONS:
Biological: Monovalent Subvirion A/H1N1 Influenza vaccine (7.5 µg of HA) — 0.5 mL, Intramuscular on Day 0 and on Day 21
  Arms: A/H1N1 Vaccine Group 1
Biological: Monovalent Subvirion A/H1N1 Influenza vaccine (15 µg of HA) — 0.5 mL, Intramuscular on Day 0 and Day 21
  Arms: A/H1N1 Vaccine Group 2
Biological: Monovalent Subvirion A/H1N1 Influenza vaccine (30 µg of HA) — 0.5 mL, Intramuscular on Day 0 and day 21
  Arms: A/H1N1 Vaccine Group 3
Biological: Normal saline solution (placebo) — 0.5 mL, Intramuscular on Day 0 and Day 21
  Arms: Placebo Group

SUMMARY:
The purpose of the study is to evaluate different doses of the Influenza A/H1N1 pandemic vaccine.

Primary Objectives:

* To describe the immunogenicity of the candidate vaccines after each injection.
* To describe the safety of the candidate vaccines after each injection.

DETAILED DESCRIPTION:
Participants will receive two injections of their randomized vaccine on Day 0 and Day 21, respectively.

ELIGIBILITY:
Inclusion Criteria :

* Healthy adults aged 18 years or older on the day of inclusion
* Informed consent has been signed and dated
* Able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination, until at least 4 weeks after last vaccination.

Exclusion Criteria :

* Known pregnancy or positive urine pregnancy test
* Currently breastfeeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months which might interfere with the assessment of immune response
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B antigen, or Hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Self reported thrombocytopenia contraindicating intramuscular (IM) vaccination
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Chronic illness that in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator.
* Previous participation in a swine-origin H1N1 pandemic flu trial except if performed in 1976
* Any confirmed case of influenza (including swine-origin A/H1N1 Influenza) since March 2009
* Febrile illness (temperature ≥ 100.4°F [≥ 38.0°C]) or moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination
* Personal or family history of Guillain-Barré syndrome
* Active neoplastic disease or a history of any hematologic malignancy
* Known seizure/epilepsy history and/or taking anti-seizure medication
* Receipt of psychiatric drugs. Subjects receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without decompensating symptoms will be allowed to enroll in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (15):
- United States (15):
  - Hoover, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - South Miami, Florida
  - Maddisonville, Kentucky
  - Springfield, Missouri
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mt. Pleasant, South Carolina
  - Knoxville, Tennessee
  - Austin, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia

REFERENCES:
- [Result] Plennevaux E, Sheldon E, Blatter M, Reeves-Hoche MK, Denis M. Immune response after a single vaccination against 2009 influenza A H1N1 in USA: a preliminary report of two randomised controlled phase 2 trials. Lancet. 2010 Jan 2;375(9708):41-8. doi: 10.1016/S0140-6736(09)62026-2. Epub 2009 Dec 15. PMID 20018365
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 06 August 2009 to 07 August 2009 at 15 US clinical centers.
Pre-assignment Details: A total of 849 participants who met the inclusion and exclusion criteria were enrolled, vaccinated, and included in data analysis.
Groups:
- A/H1N1 Vaccine Group 1: Participants who received a dose of A/H1N1 vaccine (7.5 µg hemagglutinin) intramuscularly on Day 1 and Day 21, respectively.
- A/H1N1 Vaccine Group 2: Participants who received a dose of A/H1N1 Vaccine (15 µg hemagglutinin) intramuscularly, on Day 1 and Day 21, respectively.
- A/H1N1 Vaccine Group 3: Participants who received a dose of A/H1N1 Vaccine (30 µg hemagglutinin) intramuscularly on Day 1 and Day 21, respectively.
- Placebo Group: Participants who received a dose of placebo (saline) intramuscularly on Day 1 and Day 21, respectively.
Period: Overall Study
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Started | 249 | 254 | 247 | 99
Completed | 227 | 239 | 233 | 91
Not Completed | 22 | 15 | 14 | 8
Not completed — Adverse Event | 2 | 0 | 1 | 2
Not completed — Protocol Violation | 18 | 10 | 11 | 6
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group | Total
Number analyzed (Participants) | 249 | 254 | 247 | 99 | 849
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 150 | 152 | 148 | 49 | 499
  >=65 years | 99 | 102 | 99 | 50 | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (19.2) | 53.4 (18.9) | 54.4 (18.4) | 56.4 (18.1) | 53.4 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 143 | 145 | 57 | 485
  Male | 109 | 111 | 102 | 42 | 364
Region of Enrollment [Number; unit: participants]
  United States | 249 | 254 | 247 | 99 | 849

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antibody Titers ≥ 10 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age 18 to 64 Years
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and day 21 post-vaccination
Population: Pre- and post-vaccination antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 124 | 128 | 132 | 45
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 10 | 69 | 70 | 61 | 23
  Post-Vaccination 1 (Day 21) Titers at ≥ 10 | 124 | 127 | 132 | 21
  Post-Vaccination 2 (Day 42) Titers at ≥ 10 | 124 | 128 | 132 | 22

2. Primary Outcome: Number of Participants With Antibody Titers ≥ 40 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age 18 to 64 Years
Description: Seroprotection: Antibody titer ≥ 40 1/dil. Antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and Day 21 post-vaccination
Population: Antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 124 | 128 | 132 | 45
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 40 | 27 | 37 | 32 | 11
  Post-Vaccination 1 (Day 21) Titers at ≥ 40 | 118 | 126 | 132 | 10
  Post-Vaccination 2 (Day 42) Titers at ≥ 40 | 124 | 127 | 131 | 11

3. Primary Outcome: Geometric Mean Titers (GMT) of Antibodies Against A/California (H1N1 Vaccine) Strain - Age 18 to 64 Years
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Antibody titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 124 | 128 | 132 | 45
Titers
  Pre-Vaccination 1 (Day 0) GMT | 14.5 [11.6 to 18.1] | 17.3 [13.5 to 22.1] | 14.1 [11.0 to 18.0] | 14.0 [9.31 to 21.2]
  Post-Vaccination 1 (Day 21) GMT | 708 [555 to 903] | 1362 [1073 to 1729] | 1526 [1229 to 1895] | 13.1 [8.89 to 19.3]
  Post-Vaccination 2 (Day 42) GMT | 800 [650 to 986] | 1329 [1059 to 1669] | 1331 [1082 to 1638] | 13.5 [9.23 to 19.8]

4. Primary Outcome: Number of Participants With Antibody Titers ≥ 10 1/Dilution (1/Dil) Against A/California (H1N1) Strain - Age ≥ 65 Years
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Pre- and post-vaccination antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 87 | 87 | 85 | 39
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 10 | 64 | 54 | 60 | 24
  Post-Vaccination 1 (Day 21) Titers at ≥ 10 | 87 | 87 | 85 | 23
  Post-Vaccination 2 (Day 42) Titers at ≥ 10 | 87 | 87 | 85 | 26

5. Primary Outcome: Number of Participants With Antibody Titers ≥ 40 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age ≥ 65 Years
Description: as for outcome 2
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Pre- and post-vaccination antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 87 | 87 | 85 | 39
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 40 | 21 | 21 | 24 | 10
  Post-Vaccination 1 (Day 21) Titers at ≥ 40 | 82 | 80 | 80 | 9
  Post-Vaccination 2 (Day 42) Titers at ≥ 40 | 85 | 83 | 85 | 10

6. Primary Outcome: Geometric Mean Titers (GMT) of Antibodies Against A/California (H1N1 Vaccine) Strain - Age ≥ 65 Years
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Antibody titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 87 | 87 | 85 | 39
Titers
  Pre-Vaccination 1 (Day 0) GMT | 19.1 [14.8 to 24.5] | 14.7 [12.0 to 18.1] | 18.3 [14.1 to 23.7] | 17.5 [11.0 to 27.9]
  Post-Vaccination 1 (Day 21) GMT | 319 [229 to 443] | 423 [298 to 600] | 578 [408 to 819] | 17.5 [11.2 to 27.4]
  Post-Vaccination 2 (Day 42) GMT | 359 [268 to 481] | 416 [311 to 556] | 604 [442 to 827] | 19.0 [12.1 to 29.7]

7. Primary Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction - Age 18 to 64 Years
Description: Solicited Injection Site Reactions: Pain, erythema (redness), swelling, induration (hardening), ecchymosis (bruising). Solicited systemic reactions: Fever (temperature), headache, malaise (feeling unwell), myalgia (muscle aches and pains), shivering (chills).
Time Frame: Days 0 to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 149 | 152 | 149 | 49
Participants
  Any Solicited Injection Site Reaction - Any Dose | 65 | 60 | 73 | 9
  Grade 3 Injection Site Reaction - Any Dose | 4 | 1 | 2 | 0
  Any Pain - Post Dose 1 | 53 | 43 | 48 | 8
  Any Pain - Post Dose 2 | 39 | 42 | 56 | 4
  Any Pain - Any Dose | 64 | 59 | 72 | 9
  Grade 3 Pain (Prevents daily activity) - Any Dose | 4 | 1 | 2 | 0
  Any Erythema - Post Dose 1 | 0 | 0 | 0 | 0
  Any Erythema - Post Dose 2 | 0 | 0 | 2 | 0
  Any Erythema - Any Dose | 0 | 0 | 2 | 0
  Grade 3 Erythema (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Swelling - Post Dose 1 | 1 | 2 | 2 | 0
  Any Swelling - Post Dose 2 | 0 | 2 | 2 | 0
  Any Swelling - Any Dose | 1 | 3 | 3 | 0
  Grade 3 Swelling (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Induration - Post Dose 1 | 1 | 1 | 1 | 0
  Any Induration - Post Dose 2 | 0 | 2 | 2 | 0
  Any Induration - Any Dose | 1 | 2 | 2 | 0
  Grade 3 Induration (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Ecchymosis - Post Dose 1 | 1 | 1 | 0 | 0
  Any Ecchymosis - Post Dose 2 | 1 | 1 | 1 | 0
  Any Ecchymosis - Any Dose | 2 | 1 | 1 | 0
  Grade 3 Ecchymosis (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Solicited Systemic Reaction - Any Dose | 81 | 73 | 78 | 24
  Any Grade 3 Solicited Systemic Reaction - Any Dose | 10 | 6 | 3 | 4
  Any Fever - Post Dose 1 | 1 | 1 | 2 | 1
  Any Fever - Post Dose 2 | 1 | 0 | 1 | 0
  Any Fever - Any Dose | 2 | 1 | 2 | 1
  Grade 3 Fever (≥ 102.1 F or ≥ 39.0 C) - Any Dose | 1 | 0 | 0 | 1
  Any Headache - Post Dose 1 | 48 | 48 | 40 | 16
  Any Headache - Post Dose 2 | 36 | 21 | 31 | 11
  Any Headache - Any Dose | 60 | 55 | 53 | 19
  Grd 3 Headache (Prevents daily activity), Any Dose | 5 | 5 | 2 | 3
  Any Malaise - Post Dose 1 | 34 | 23 | 27 | 9
  Any Malaise - Post Dose 2 | 22 | 15 | 25 | 6
  Any Malaise - Any Dose | 43 | 31 | 42 | 13
  Grd 3 Malaise (Prevents daily activity) - Any Dose | 6 | 3 | 2 | 2
  Any Myalgia - Post Dose 1 | 43 | 30 | 33 | 11
  Any Myalgia - Post Dose 2 | 22 | 16 | 26 | 5
  Any Myalgia - Any Dose | 49 | 34 | 49 | 13
  Grd 3 Myalgia (Prevents daily activity) - Any Dose | 6 | 2 | 0 | 2
  Any Shivering - Post Dose 1 | 10 | 2 | 8 | 2
  Any Shivering - Post Dose 2 | 2 | 0 | 3 | 0
  Any Shivering - Any Dose | 12 | 2 | 9 | 2
  Grade 3 Shivering (Prevents activity) - Any Dose | 1 | 0 | 0 | 1

8. Primary Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction - Age ≥ 65 Years
Description: as for outcome 7
Time Frame: Days 0 to 7 post-vaccination
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Number analyzed (Participants) | 99 | 102 | 99 | 50
Participants
  Any Solicited Injection Site Reaction - Any Dose | 20 | 19 | 27 | 2
  Grade 3 Injection Site Reaction - Any Dose | 0 | 0 | 1 | 0
  Any Pain - Post Dose 1 | 10 | 12 | 16 | 0
  Any Pain - Post Dose 2 | 10 | 14 | 16 | 2
  Any Pain - Any Dose | 18 | 19 | 24 | 2
  Grade 3 Pain (Prevents daily activity) - Any Dose | 0 | 0 | 1 | 0
  Any Erythema - Post Dose 1 | 1 | 0 | 1 | 0
  Any Erythema - Post Dose 2 | 1 | 0 | 2 | 0
  Any Erythema - Any Dose | 2 | 0 | 3 | 0
  Grade 3 Erythema (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Swelling - Post Dose 1 | 0 | 0 | 2 | 0
  Any Swelling - Post Dose 2 | 0 | 0 | 2 | 1
  Any Swelling - Any Dose | 0 | 0 | 3 | 1
  Grade 3 Swelling (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Induration - Post Dose 1 | 0 | 0 | 0 | 0
  Any Induration - Post Dose 2 | 0 | 1 | 0 | 0
  Any Induration - Any Dose | 0 | 1 | 0 | 0
  Grade 3 Induration (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Ecchymosis - Post Dose 1 | 2 | 0 | 2 | 0
  Any Ecchymosis - Post Dose 2 | 0 | 1 | 0 | 1
  Any Ecchymosis - Any Dose | 2 | 1 | 2 | 1
  Grade 3 Ecchymosis (> 10 cm) - Any Dose | 0 | 0 | 0 | 0
  Any Solicited Systemic Reaction - Any Dose | 28 | 22 | 32 | 13
  Any Grade 3 Solicited Systemic Reaction - Any Dose | 2 | 1 | 1 | 0
  Any Fever - Post Dose 1 | 0 | 0 | 1 | 1
  Any Fever - Post Dose 2 | 0 | 0 | 0 | 1
  Any Fever - Any Dose | 0 | 0 | 1 | 2
  Grade 3 Fever (≥ 102.1 ºF or ≥ 39.0 ºC) - Any Dose | 0 | 0 | 0 | 0
  Any Headache - Post Dose 1 | 11 | 10 | 16 | 6
  Any Headache - Post Dose 2 | 9 | 7 | 8 | 9
  Any Headache - Any Dose | 16 | 13 | 21 | 11
  Grd 3 Headache (Prevents daily activity), Any Dose | 1 | 0 | 0 | 0
  Any Malaise - Post Dose 1 | 4 | 7 | 15 | 4
  Any Malaise - Post Dose 2 | 11 | 4 | 7 | 5
  Any Malaise - Any Dose | 14 | 9 | 21 | 8
  Grd 3 Malaise (Prevents daily activity) - Any Dose | 1 | 0 | 1 | 0
  Any Myalgia - Post Dose 1 | 7 | 9 | 11 | 2
  Any Myalgia - Post Dose 2 | 5 | 10 | 8 | 5
  Any Myalgia - Any Dose | 11 | 16 | 17 | 6
  Grd 3 Myalgia (Prevents daily activity) - Any Dose | 1 | 1 | 1 | 0
  Any Shivering - Post Dose 1 | 1 | 0 | 2 | 1
  Any Shivering - Post Dose 2 | 2 | 3 | 0 | 2
  Any Shivering - Any Dose | 3 | 3 | 2 | 3
  Grade 3 Shivering (Prevents activity) - Any Dose | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to up to 6 months post-vaccination 2.
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | A/H1N1 Vaccine Group 3 | Placebo Group
Serious Adverse Events (participants affected / at risk) | 8/248 | 7/254 | 7/248 | 4/99
Other Adverse Events (participants affected / at risk) | 82/248 | 78/254 | 96/248 | 30/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/H1N1 Vaccine Group 1 (N=248) | A/H1N1 Vaccine Group 2 (N=254) | A/H1N1 Vaccine Group 3 (N=248) | Placebo Group (N=99)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignan (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Non-Hodgkins lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Global amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | A/H1N1 Vaccine Group 1 (N=248) | A/H1N1 Vaccine Group 2 (N=254) | A/H1N1 Vaccine Group 3 (N=248) | Placebo Group (N=99)
Injection site pain (General disorders) | 82/242 | 78/249 | 96/246 | 11/98
Headache (Nervous system disorders) | 76/242 | 68/249 | 74/246 | 30
Malaise (General disorders) | 57/242 | 40/249 | 63/246 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 60/242 | 50/249 | 66/246 | 19
Shivering (General disorders) | 15/242 | 15/249 | 11/246 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications